CLINICAL TRIAL: NCT06620887
Title: SICKLE CELL DISEASE AND PREGNANCY : HEMAGO Monitoring and Impact on the Occurrence of Maternal, Obstetrics and Perinatal Complications in Sickle Cell Patients
Brief Title: HEMAGO Monitoring and Impact on the Occurrence of Complications During Pregnancy in Sickle Cell Patients
Acronym: HEMAGO
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 24-5120
Record Dates: First submitted 2024-09-27; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Sickle Cell Disease and Pregnancy
Keywords: Sickle cell disease ; genetic disease ; anemia ; pregnancy ; obstetrics complications
MeSH Terms: conditions — Anemia, Sickle Cell; Genetic Diseases, Inborn; Anemia | interventions — Mortality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnancies before HEMAGO: Pregnancies follow-up before HEMAGO : complications and outcomes of pregnancies in sickle cell patients which had a classical follow-up.
  Interventions: Other: Evaluate the impact of HEMAGO program on maternal morbidity and mortality in sickle cell disease patients during their pregnancies.
- Pregnancies HEMAGO following-up: Pregnancies in sickle cell patients follow-up by HEMAGO : complications and outcomes of pregnancies in sickle cell disease patients which were monitored by HEMAGO program.
  Interventions: Other: Evaluate the impact of HEMAGO program on maternal morbidity and mortality in sickle cell disease patients during their pregnancies.

INTERVENTIONS:
Other: Evaluate the impact of HEMAGO program on maternal morbidity and mortality in sickle cell disease patients during their pregnancies. — HEMAGO pregnancy monitoring is a joint consultation program between the sickle cell disease hematologist and an obstetrician. This program was implemented in April 2016 at the Croix-Rousse maternity Hospital. This program offers close, complete and personalized pregnancy monitoring for each patient with major sickle cell syndrome.
  These are follow-up consultations once a month until 24 weeks then every 15 days until delivery. At each consultation, doctors evaluate a general and obstetric clinical examination. The team establishes a precise schedule adapted to each patient for pregnancy monitoring : monthly blood tests, monthly ultrasounds with maternal and fetal Doppler, adaptation of basic treatment, transfusion exchange program according to eligibility criteria, and organization of childbirth.

SUMMARY:
Sickle cell disease is the most common monosemic genetic disease in the world and affects approximately 32,000 people in France. In recent years, improvements in the management of this pathology have led to a steady increase in the life expectancy of sickle cell patients.

Women with sickle cell disease are increasingly likely to have one or more pregnancies.

Several studies have shown that these pregnancies are marked by maternal morbidity due to acute sickling crises, thromboembolism, infection, chronic end-organ dysfunction, or pre-eclampsia (PE), while neonatal outcomes may be intrauterine growth retardation (IUGR), preterm delivery, small infants for gestational age, stillbirth, and neonatal death.

Consequently, monitoring pregnancies in sickle cell patients represents a complex medical challenge due to the risk of potentially serious maternal and fetal complications. Multidisciplinary follow-up is then crucial to monitor and manage these possible complications.

The double hematologist-obstetrician consultation program (HEMAGO) offers complete and adapted close follow-up, in order to minimize the risks for the mother and the unborn child.

This study aims to evaluate the impact of this HEMAGO monitoring on the various maternal and obstetric complications by comparing the outcome of pregnancies of patients who were followed before the implementation of this device to patients who were followed in the frame their pregnancy through this program.

ELIGIBILITY:
Inclusion Criteria:

* sickle cell disease female
* followed up for at least one pregnancy in the maternity of Croix-Rousse Hospital, Femme Mère Enfant Hospital and Lyon Sud Hospital

Exclusion Criteria:

* Minor woman

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cohort of sickle cell patients followed in the red blood cell pathology department at the Edouard Herriot Hospital and having had a pregnancy follow-up consultation in one of the three maternity wards in Lyon.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Composite criterion including in the mother : Maternal complications → Obstetrics complications → Sickle cell complications → intensive care hospitalization → death ? | These are follow-up consultations once a month until 24 weeks then every 15 days until delivery. comparing results before (January 2005 to March 2016) and after HEMAGO (April 2016 - February 29, 2024)
  Maternal complications :
  * Obstetrics complications : pre-eclampsia or Hellp syndrome / intra-uterine growth restriction (IUGR) / preterm labor / chorioamniotis / intrauterine death
  * Sickle cell complications (vaso-occlusive crisis (VOC) / acute chest syndrome / cerebral stroke)
  * lung or urinary infections
  * thromboembolism
  * intensive care hospitalization
  collection of data done by rereading obstetric records by a single person.

CONTACTS AND LOCATIONS:
Overall Officials: Dr FICHEZ Axel, Dr, Principal Investigator — Service de Gynécologie-Obstétrique Hôpital de la Croix-Rousse/Groupement Hospitalier Nord
Locations (3):
- France (3):
  - Service de gynécologie-obstétrique de l'Hôpital Femme Mère Enfant, Bron
  - Croix-Rousse Hospital - Service de Gynécologie-Obstétrique, Lyon
  - Service de gynécologie-obstétrique de l'Hôpital de Lyon Sud, Lyon